CLINICAL TRIAL: NCT05007873
Title: Phase II Study Assessing Safety and Clinical Activity of the Combination of ASTX727 With Dasatinib in Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase (CML-CP)
Brief Title: ASTX727 and Dasatinib for the Treatment of Newly Diagnosed Philadelphia Chromosome or BCR-ABL Positive Chronic Myeloid Leukemia in Chronic Phase
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0271; NCI-2021-08486 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0271 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia; Philadelphia Chromosome Positive; BCR-ABL1 Positive Chronic Myelogenous Leukemia; BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dasatinib, decitabine and cedazuridine) (Experimental): Patients receive dasatinib PO QD on days 1-28. Beginning cycle 4, patients also receive decitabine and cedazuridine PO QD on days 1-3. Cycles repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive dasatinib PO QD on days 1-28. Cycles repeat every 28 days for up to 12 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Drug: Decitabine and Cedazuridine

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inqovi

SUMMARY:
This phase II trial studies the effect of ASTX727 and dasatinib in treating patients with newly diagnosed Philadelphia chromosome or BCR-ABL positive chronic myeloid leukemia in chronic phase. Philadelphia chromosome positive and BCR-ABL positive are types of genetic mutations (changes). Chemotherapy drugs, such as ASTX727, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. ASTX727 and dasatinib may help to control Philadelphia chromosome-positive chronic myeloid leukemia or BCR-ABL positive chronic myeloid leukemia in chronic phase.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the proportion of patients with previously-untreated chronic phase chronic myeloid leukemia (CML) who achieve molecular response 4 (MR4) after 6-months of the combination of decitabine and cedazuridine (ASTX727) and dasatinib 50 mg daily.

SECONDARY OBJECTIVES:

I. To estimate the proportion of patients with previously-untreated chronic phase CML who achieve MR4 after both the 3-months of the combination of ASTX727 and dasatinib 50 mg daily.

II. To estimate cumulative overall rate of molecular response 4.5 (MR4.5). III. To estimate the 12-months major molecular response (MMR) rate. IV. To estimate the proportion of patients with MR4.5 at 6-, 12-, 18-, 24-, and 36-months of therapy.

V. To estimate the proportion of patients with sustained MR4.5 of 3 years and more.

VI. To estimate the treatment-free remission rate (TFR), time to progression, and overall survival.

VII. To assess the safety of this combination.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD) on days 1-28. Beginning cycle 4, patients also receive decitabine and cedazuridine PO QD on days 1-3. Cycles repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive dasatinib PO QD on days 1-28. Cycles repeat every 28 days for up to 12 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Philadelphia chromosome (Ph)-positive or BCR-ABL positive CML in early chronic phase CML (i.e., time from diagnosis ≤12 months). Except for hydroxyurea and/or 1 to 2 doses of cytarabine patients must have received no or minimal prior therapy, defined as < 1 month (30 days) of prior Food and Drug Administration (FDA) approved tyrosine kinase inhibitor (TKI)

  * Clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph chromosome has historically been included as a criterion for accelerated phase. However, patients with clonal evolution as the only criterion of accelerated phase have a significantly better prognosis, and when present at diagnosis may not impact the prognosis at all. Thus, patients with clonal evolution at diagnosis (early disease) and no other criteria for accelerated phase will be eligible for this study.
* Eastern Cooperative Oncology Group (ECOG) performance of 0-2
* Adequate end organ function, defined as the following: total bilirubin <1.5x ULN (unless secondary to Gilbert's disease, in which case should be < 2.5x ULN), SGPT <3x ULN, creatinine clearance ≥ 30mL/min calculated using modified Crokcroft-Gault.
* Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
* Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment.

Exclusion Criteria:

* New York Heart Association (NYHA) cardiac class 3-4 heart disease
* Cardiac Symptoms: Patients meeting the following criteria are not eligible unless cleared by Cardiology:

  * Uncontrolled angina within 3 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
  * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 460 msec)
  * History of significant bleeding disorder unrelated to cancer, including unless cleared by hematologist or hemato-oncologist

    * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
    * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients with active, uncontrolled psychiatric disorders include: psychosis, major depression, and bipolar disorders
* Subject is known to be positive for human immunodeficiency virus (HIV) (HIV testing is not required)
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface [HBs] antigen negative-, anti-HBs antibody positive and anti-hepatitis B core [HBc] antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
* Women of pregnancy potential must practice an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women must continue birth control for the duration of the trial and at least 3 months after the last dose of study drug.

Pregnant or breast-feeding women are excluded.

All WOCBP must have a negative pregnancy test prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive study drug and must not be enrolled in the study

* Patients in late chronic phase (i.e., time from diagnosis to treatment > 12 months), accelerated (except as noted in inclusion criteria 4.1) or blast phase are excluded. The definitions of CML phases are as follows:

  * Early chronic phase: time from diagnosis to therapy ≤ 12 months
  * Late chronic phase: time from diagnosis to therapy > 12 months
  * Blastic phase: presence of 30% blasts or more in the peripheral blood or bone marrow
  * Accelerated phase CML: presence of any of the following features:

    * Peripheral or marrow blasts 15% or more
    * Peripheral or marrow basophils 20% or more
    * Thrombocytopenia < 100 x 10^9/L unrelated to therapy
    * Documented extramedullary blastic disease outside liver or spleen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of molecular response 4 (MR4) | At 6 months
  Will be estimated with 95% credible intervals. The association between molecular responses and demographic/ clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test.

SECONDARY OUTCOMES:
Rate of MR4.5 | At 12 months
  Will be presented with 95% confidence intervals. The association between molecular responses and demographic/ clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test.
Major molecular response rate | At 12 months
  Will be presented with 95% confidence intervals. The association between molecular responses and demographic/ clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test.
Treatment-free remission rate | Up to 15 years
  Will be presented with 95% confidence intervals. The association between molecular responses and demographic/ clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test.
Time to progression | Up to 15 years
  Survival time will be estimated using the Kaplan-Meier method. Patients who drop out of the study will be included in the time to event data as "censored data". The two-sided log-rank test will be used to assess the differences of time to events between groups.
Overall survival | Up to 15 years
  Survival time will be estimated using the Kaplan-Meier method. Patients who drop out of the study will be included in the time to event data as "censored data". The two-sided log-rank test will be used to assess the differences of time to events between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org